CLINICAL TRIAL: NCT03638102
Title: The Effect of Sleep Extension on Glucose Metabolism in Women With Previous Diagnosis of Gestational Diabetes
Brief Title: Sleep Duration in Women With Previous Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sirimon Reutrakul, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-0992
Record Dates: First submitted 2018-08-12; First posted 2018-08-20 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Gestational Diabetes
Keywords: sleep duration; glucose metabolism
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep intervention (Experimental): Sleep extension
  Interventions: Behavioral: Sleep extension
- Healthy living (Active Comparator): Health education
  Interventions: Behavioral: Healthy living

INTERVENTIONS:
Behavioral: Sleep extension — Sleep extension aims to increase sleep duration for at least 30 minutes using weekly coaching
  Arms: Sleep intervention
Behavioral: Healthy living — Participants will receive weekly health education
  Arms: Healthy living

SUMMARY:
Women with a history of gestational diabetes (GDM) are at high risk of developing diabetes in the future. Sleep disturbances are emerging as risk factors for incident diabetes. The purpose of this study is to test the effects of 6-week sleep extension in women with a history of GDM and short sleep on glucose metabolism by randomized controlled study.

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effects of a sleep extension intervention in non-diabetic women with a prior history of GDM and habitual short sleep duration on the outcomes of glucose metabolism. The participants will be randomized to a 6-week sleep extension intervention group, using technology-assisted sleep intervention, or a healthy living information control group. Glucose metabolism parameters will be assessed by an oral glucose tolerant test.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, age 18-45, with a history of GDM who currently do not have diabetes
* At least one year post-partum
* Reported habitual sleep duration <7h/night during work- or weekdays with a desire to sleep longer
* Reported time spent in bed =<8 hours
* Own a smartphone compatible with Fitbit.
* No need to provide care at night for her child(ren), defined as >3 times a week and >30 minutes at a time
* No history of obstructive sleep apnea, insomnia, or restless leg syndrome

Exclusion Criteria:

* A1C ≥6.5%
* Currently pregnant or planning pregnancy or breast feeding
* Insomnia symptoms defined as severe as assessed by the Insomnia Severity Index (score ≥15)
* Rotating shift or night shift work
* High risk for obstructive sleep apnea screened by STOP BANG questionnaire.
* Significant medical morbidities, such as congestive heart failure, cirrhosis, chronic obstructive pulmonary disease requiring oxygen, active treatment for cancer or psychiatric problem, history of stroke with neurological deficits, cognitive impairment, kidney failure requiring dialysis, illicit drug use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-diabetic women with a previous history of gestational diabetes
Enrollment: 18 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sirimon Reutrakul, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] Reutrakul S, Van Cauter E. Interactions between sleep, circadian function, and glucose metabolism: implications for risk and severity of diabetes. Ann N Y Acad Sci. 2014 Apr;1311:151-73. doi: 10.1111/nyas.12355. Epub 2014 Mar 14. PMID 24628249
- [Background] Amnakkittikul S, Chirakalwasan N, Wanitcharoenkul E, Charoensri S, Saetung S, Chanprasertyothin S, Chailurkit LO, Panburana P, Bumrungphuet S, Reutrakul S. Postpartum resolution of obstructive sleep apnea in women with gestational diabetes and the relationship with glucose metabolism. Acta Diabetol. 2018 Jul;55(7):751-754. doi: 10.1007/s00592-018-1127-x. Epub 2018 Mar 15. No abstract available. PMID 29546578
- [Background] Baron KG, Duffecy J, Reid K, Begale M, Caccamo L. Technology-Assisted Behavioral Intervention to Extend Sleep Duration: Development and Design of the Sleep Bunny Mobile App. JMIR Ment Health. 2018 Jan 10;5(1):e3. doi: 10.2196/mental.8634. PMID 29321122
- [Background] Mohr DC, Duffecy J, Ho J, Kwasny M, Cai X, Burns MN, Begale M. A randomized controlled trial evaluating a manualized TeleCoaching protocol for improving adherence to a web-based intervention for the treatment of depression. PLoS One. 2013 Aug 21;8(8):e70086. doi: 10.1371/journal.pone.0070086. eCollection 2013. PMID 23990896
- [Derived] Reutrakul S, Martyn-Nemeth P, Quinn L, Rydzon B, Priyadarshini M, Danielson KK, Baron KG, Duffecy J. Effects of Sleep-Extend on glucose metabolism in women with a history of gestational diabetes: a pilot randomized trial. Pilot Feasibility Stud. 2022 Jun 4;8(1):119. doi: 10.1186/s40814-022-01076-2. PMID 35659776

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sleep Intervention | Healthy Living
Started | 12 | 6
Completed | 9 | 5
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Intervention | Healthy Living | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (2.6) | 38.7 (6) | 40.8 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 15
Sleep duration [Mean (Standard Deviation); unit: minutes] — Population: one person dropped out
  minutes
    number analyzed (Participants) | 12 | 5 | 17
    (all) | 369 (31) | 408 (90) | 383 (33)
fasting glucose [Mean (Standard Deviation); unit: mg/dL] — Population: one person dropped out
  mg/dL
    number analyzed (Participants) | 12 | 5 | 17
    (all) | 102.3 (12.9) | 96.4 (3.8) | 100.2 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Fasting Glucose
Description: Changes in fasting glucose between baseline and 6 weeks
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Living | Sleep Intervention
Number analyzed (Participants) | 5 | 9
mg/dL | 10.4 (8.2) | 1.6 (9.4)

2. Primary Outcome: Sleep Duration Change
Description: Changes in sleep duration from baseline to 6 weeks
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Healthy Living | Sleep Intervention
Number analyzed (Participants) | 5 | 9
minutes | -9.1 (20.4) | 26.9 (42.5)

3. Secondary Outcome: HOMA-IR Change
Description: HOMA-IR change at week 0 to week 6. This is an index of fasting insulin resistance, and the higher reflects greater insulin resistance. Generally, a value greater than 2 is suggestive of insulin resistance
Time Frame: baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sleep Intervention | Healthy Living
Number analyzed (Participants) | 9 | 5
index | 0.7 (1.4) | 0.59 (1.08)

4. Secondary Outcome: Change in Subjective Sleep Quality
Description: Pittsburgh sleep quality index (range 0 to 21 with higher score reflecting worse sleep quality)
Time Frame: Baseline and week 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Healthy Living | Sleep Intervention
Number analyzed (Participants) | 5 | 9
Score on a scale | -2.0 (4.2) | -2.8 (3.2)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Healthy Living | Sleep Intervention
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03638102/Prot_SAP_000.pdf